CLINICAL TRIAL: NCT05326542
Title: ESWL Combined With ERCP and Laser Lithotripsy Combined With ERCP In Treatment of Pancreatic Duct Stones With Chronic Pancreatitis: a Randomized Controlled Trial
Brief Title: Comparison of Efficacy of ESWL and Laser Lithotripsy in Chronic Pancreatitis With ERCP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Professor, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ECLIPSE20220312
Record Dates: First submitted 2022-04-06; First posted 2022-04-13 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Pancreatitis, Chronic; Pancreatic Duct Stone
Keywords: Cholangiopancreatography, Endoscopic Retrograde; Lithotripsy
MeSH Terms: conditions — Pancreatitis, Chronic | interventions — Lithotripsy; Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESWL and ERCP (Experimental): The patients will receive intravenous analgesia (flurbiprofen and remifentanil) before the ESWL (Compact Delta II; Dornier Med Tech, Wessling, Germany). The time scale between the last ESWL session and following ERCP will be greater than 48h. ERCP will be performed under conscious sedation with intramuscular administration of diazepam 2.5-5.0 mg and pethidine 25-50 mg. If necessary, endoscopic sphincterotomy will be performed. A dilating bougie or balloon will be used to dilate the stenosis after sphincterotomy. Standard techniques (i.e., extraction basket, extraction balloon, or both) will be used for stone removal. A pancreatic duct stent or a nasopancreatic catheter will be inserted for temporary drainage if necessary.
  Interventions: Procedure: ESWL and ERCP
- LL and ERCP (Active Comparator): ERCP will be performed under conscious sedation with intramuscular administration of diazepam 2.5-5.0 mg and pethidine 25-50 mg. If necessary, endoscopic sphincterotomy will be performed. A dilating bougie or balloon will be used to dilate the stenosis after sphincterotomy. After that, laser lithotripsy will be performed. Standard techniques (i.e., extraction basket, extraction balloon, or both) will be used for stone removal. A pancreatic duct stent or a nasopancreatic catheter will be inserted for temporary drainage if necessary.
  Interventions: Procedure: LL and ERCP

INTERVENTIONS:
Procedure: ESWL and ERCP — First, ESWL will be used for lithotripsy, and then ERCP will be performed to clear the stones after lithotripsy.
  Arms: ESWL and ERCP
Procedure: LL and ERCP — After establishing the working channel under ERCP, the stone will be crushed with a laser lithotripter, and then ERCP will clear the stones after lithotripsy.
  Arms: LL and ERCP

SUMMARY:
This study will compare the efficacy of ESWL and Laser Lithotripsy in the treatment of pancreatic duct stones with ERCP.

DETAILED DESCRIPTION:
Chronic pancreatitis (CP) is an inflammatory disease that can causes progressive fibrosis of pancreatic tissue and eventually leads to damage of pancreatic exocrine and endocrine. According to statistics, the prevalence of CP in China is 13/10 million, which is still increasing. Pancreatic duct stones are the most important pathological changes of CP. More than 50% of patients with CP are accompanied by pancreatic duct stones, which can lead to pancreatic duct obstruction, hypertension and tissue ischemia. Removal of pancreatic duct stones under Endoscopic Retrograde Cholangiopancreatography (ERCP) are the first choice. ERCP is effective in the treatment of pancreatic duct stones by using basket and/or balloon catheter. But in most cases, ERCP is only suitable for the treatment of pancreatic duct stones (diameter < 5mm) located in the head/body of the Pancreatic Duct (PD). PD stones larger than 5mm generally require Extracorporeal Shock Wave Lithotripsy (ESWL) or Endoscopic Intraductal Lithotripsy (EIL) for pretreatment. EIL includes Electrohydraulic Lithotripsy (EHL) and Laser Lithotripsy (LL).

ESWL first locates the stone by X-ray, and then uses an electromagnetic pulse generator to direct a higher-energy shock wave to the stone, so that the stone is crushed by thousands of shock waves. The principle of laser lithotripsy is to make the stone absorb strong infrared rays and generate shock waves to achieve the purpose of fragmenting the stone.

In view of the fact that there is no relevant research comparing the overall efficacy of ESWL combined with ERCP and EIL combined with ERCP, it is necessary to evaluate the differences in the therapeutic effects and complications of the two for PD stones. This research helps to provide evidence-based medical evidence, guide physicians' clinical practice, improve the quality of patients' lives, and reduce the economic burden of patients.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic adult patients diagnosed with chronic pancreatitis and pancreatic duct stones;
* at least one stone (>5 mm in diameter) located in the pancreatic duct of the head/body of the pancreas;
* dilation of the proximal pancreatic duct.

Exclusion Criteria:

* history of ERCP or ESWL treatment;
* suspected to have malignant tumors;
* history of pancreatic surgery or gastrojejunostomy (Billroth II);
* pancreatic pseudocyst with a diameter >4cm;
* bile duct stricture secondary to cholangitis or chronic pancreatitis;
* acute pancreatitis exacerbation or acute exacerbation of chronic pancreatitis (including biliary pancreatitis);
* coagulation dysfunction (INR≥1.5 or platelet count≤50×10^9/L);
* pregnant or breastfeeding women;
* patients who refused to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
technical success rates | during ERCP procedure
  Technical success rates refer to the successful completion of standard procedures or the occurrence of complete spontaneous stone removal.
clearance rates of pancreatic duct stones | during ERCP procedure
  Clearance rates have been defined as complete, partial, or failure if the proportion of stones cleared was > 90%, 50% - 90%, or < 50%, respectively.

SECONDARY OUTCOMES:
time taken to completely clear the stone | during ESWL and ERCP procedure
  The time taken to completely clear the stones.
postoperative complications | 30 days after ERCP procedure
  Major post-ERCP complications includes post-ERCP pancreatitis, bleeding, infection, and perforation, which are classified as mild, moderate, or severe, depending mainly on the length of hospitalization and the need for invasive treatment.
success rates of pancreatic duct decompression | during ERCP procedure
  Successful removal of pancreatic duct obstruction factors by clearing stones and/or placing pancreatic duct stents/nasopancreatic catheters.

OTHER OUTCOMES:
abdominal pain relief rate | 30 days after ERCP procedure
  Postoperative and preoperative abdominal pain was assessed using the Visual Analogue Scale (VAS). VAS can be calculated ranging from 0 (no pain) to 100 (severe pain).

CONTACTS AND LOCATIONS:
Overall Officials: Liang-hao Hu, MD, Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hao L, Liu Y, Xie T, Wang T, Guo HL, Pan J, Wang D, Bi YW, Ji JT, Xin L, Du TT, Lin JH, Zhang D, Zeng XP, Zou WB, Chen H, Li BR, Liao Z, Cong ZJ, Shi RH, Li ZS, Hu LH. Risk Factors and Nomogram for Pancreatic Stone Formation in Chronic Pancreatitis over a Long-Term Course: A Cohort of 2,153 Patients. Digestion. 2020;101(4):473-483. doi: 10.1159/000500941. Epub 2019 Jun 25. PMID 31238312